CLINICAL TRIAL: NCT07094347
Title: Effects of Intradialytic Inspiratory Muscle Training on Functional Capacity in Hemodialysis Patients
Acronym: Hemodialysis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KA24/416
Record Dates: First submitted 2025-05-28; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Hemodialysis
Keywords: powerbreathe

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory Muscle Training Group (Experimental): The individuals in the study group will be given a 12-week respiratory muscle training after the first assessment and training session. The Powerbreathe® threshold resistance loading device (POWERbreathe, HaB International) will be used for this training program that strengthens the inspiratory muscles. The PowerBreathe® device is a threshold device that creates resistance to inspiration. This resistance is created by the spring tension in the device's mechanism. The device has a mechanism that is adjusted according to 9 different levels in its mechanism specific to the individuals using it.
  Interventions: Device: inspiratory muscle training
- control (No Intervention): At the beginning of the study after the first assessment, the control group will be given a training session lasting approximately 30 minutes. During the training session, participants will be given training on bronchial hygiene techniques and respiratory control, pursed lip breathing, diaphragmatic breathing exercises and thoracic expansion exercises that will improve lung health. Individuals in the control group will only receive the training session after the assessment.

INTERVENTIONS:
Device: inspiratory muscle training — Powerbreathe® threshold resistance loading device (POWERbreathe, HaB International) will be used for this training program that strengthens the inspiratory muscles. The PowerBreathe® device is a threshold device that creates resistance to inspiration. This resistance is created by the spring tension in the device mechanism. The device has a mechanism that is adjusted according to 9 different levels in its mechanism specific to the individuals using it.
  Arms: Inspiratory Muscle Training Group

SUMMARY:
There is a need for long-term sustainable studies that will increase the potential health benefits in hemodialysis patients. Inspiratory muscle training, one of the recommended treatments to increase exercise capacity and quality of life during dialysis treatment in people with chronic renal failure, is a method that can be applied intradialytically, in addition to being easy to apply, cheap and sustainable. It improves functional capacity by increasing respiratory muscle strength. In this context, our study aims to investigate the effects of inspiratory muscle training on functional parameters and on hemodialysis patients with a personalized portable device and to add it to the literature.

DETAILED DESCRIPTION:
Chronic kidney disease is defined as abnormalities in kidney structure or function that have been present for more than three months and will adversely affect health. Two markers used to define chronic kidney disease, which is characterized by progressive loss of kidney mass and function, are glomerular filtration rate (GFR) and albumin-creatinine ratio. Chronic kidney disease can be divided into five stages according to GFR, and the most severe end-stage chronic kidney disease is also defined as chronic renal failure and requires renal replacement therapy to maintain homeostasis. The most commonly applied method of renal replacement in our country is hemodialysis.

It is known that muscle atrophy, where muscle regeneration and repair capacity decrease, is frequently seen in chronic kidney disease patients. Although it is partly due to aging, muscle atrophy is frequently seen due to the accumulation of uremic toxins, inflammation, insulin resistance, malnutrition and lack of physical activity; increased muscle loss also increases the risk of morbidity, mortality and end-stage renal disease in patients.

Studies have shown that there is a decrease in respiratory muscle strength as well as skeletal muscle strength in chronic kidney disease patients. Decreased respiratory muscle strength causes individuals to have low cardiorespiratory fitness, and chronic kidney disease patients face limitations in daily life activities and increased mortality.

Pulmonary system involvement and decreased exercise tolerance are among the important causes of functional capacity and disease-related complications in chronic kidney disease patients. Inspiratory muscle strength is related to functional capacity in hemodialysis patients. In the literature, it is shown that inspiratory muscle training improves functional parameters and modulates inflammatory biomarkers, as in aerobic and combined exercise training. Inspiratory muscle training is a useful method to increase peripheral and inspiratory muscle strength, respiratory function, quality of life and balance, and to reduce dyspnea and fatigue in patients with chronic kidney disease.

Exercises performed during dialysis are called intradialytic exercises. It does not require extra time to exercise; The advantages of this exercise protocol include the fact that patients can be monitored by healthcare professionals during exercise and that any complications can be detected and treated immediately, and that intradialytic exercise increases blood flow to the muscles and increases solute removal. Inspiratory muscle training, one of the recommended treatments to increase exercise capacity and quality of life during dialysis treatment in people with chronic renal failure, is a method that can be applied intradialytically, in addition to being easy to apply, cheap and sustainable. It improves functional capacity by increasing respiratory muscle strength. It is stated that inspiratory muscle training protocols applied in the range of 30-60% of the individual's maximum inspiratory pressure improve respiratory muscle strength, functional capacity and quality of life in patients with chronic renal failure. However, the number of studies showing the effects of this type of training applied at different intensities in dialysis patients is quite low. In addition, the effects of intradialytic inspiratory muscle training applications have not yet been shown. There is a need for long-term sustainable studies in the literature that will increase the potential health benefits in hemodialysis patients. In this context, our study aims to investigate the effects of inspiratory muscle training on functional parameters and its contribution to the literature with a personalized portable device in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Being on hemodialysis for at least 6 months
* Being on hemodialysis for 4 hours, 3 days a week
* Not having had a transplant
* Being able to continue sitting and standing
* Being able to walk without assistance
* Being willing to participate in the study

Exclusion Criteria:

* Individuals with communication and/or cognitive problems that are unable to fulfill the assessment and treatment requirements
* Patients with uncontrolled cardiac, pulmonary or other systemic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Inspiratory muscle strength | The individuals participating in the study will be evaluated twice: before the application (week 0) and after the application (after 12 weeks).
  The respiratory muscle strength measuring device Power Breathe (Power Breathe, K5, HaB International Ltd England) will be used to assess inspiratory muscle strength. During the assessment, the patient will be asked to sit in a chair with back support and no arm support, with shoulders relaxed, and a nose clip will be used. Patients will be asked to take a deep breath through the device placed in their mouth. The inspiratory force index (S-index) obtained as a result of the measurement will be recorded.

SECONDARY OUTCOMES:
Exercise Capacity Assessment | The individuals participating in the study will be evaluated twice: before the application (week 0) and after the application (after 12 weeks).
  The 6-minute walk test (6MWT), which is clinically easy to apply and reliable, will be used to assess the functional capacity of individuals.The 6-minute walk test (6MWT), which is clinically easy to apply and reliable, will be used to assess the functional capacity of individuals. At the end of 6 minutes, the distance walked in meters (m) will be recorded.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Katayifci N, Huzmeli I, Iri S D, Turgut FH. Effects of different inspiratory muscle training protocols on functional exercise capacity and respiratory and peripheral muscle strength in patients with chronic kidney disease: a randomized study. BMC Nephrol. 2024 May 29;25(1):184. doi: 10.1186/s12882-024-03610-1. PMID 38811888